CLINICAL TRIAL: NCT05351593
Title: A Phase I/II Study of Tafasitamab Plus Lenalidomide in Relapsed CNS Lymphoma
Brief Title: Tafasitamab Plus Lenalidomide in Relapsed CNS Lymphoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: James Rubenstein (Other)
Collaborators: Incyte Corporation (Industry)
Responsible Party: Sponsor-Investigator, James Rubenstein, Principal Investigator, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 212531; NCI-2022-03704 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2022-04-22; First posted 2022-04-28 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: CNS Lymphoma; Primary Central Nervous System Lymphoma; Secondary Central Nervous System Lymphoma
MeSH Terms: interventions — tafasitamab; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Phase 1 (Tafasitamab, Lenalidomide) (Experimental): Participants will be given 12mg of Tafasitamab on days 1, 4, 8, 15, and 22 of cycle 1, days 1, 8, 15, and 22 of cycles 2 & 3, and days 1 and 15 for any cycle thereafter. Participants will also be given daily Lenalidomide on days 1-21 of each cycle.
  Interventions: Drug: Tafasitamab; Drug: Lenalidomide
- Phase 2 (Tafasitamab, Lenalidomide) (Experimental): Participants will be given 12mg of Tafasitamab on days 1, 4, 8, 15, and 22 of cycle 1, days 1, 8, 15, and 22 of cycles 2 & 3, and days 1 and 15 for any cycle thereafter. Participants will also be given daily Lenalidomide on days 1-21 of each cycle at the recommended phase 2 dose.
  Interventions: Drug: Tafasitamab; Drug: Lenalidomide

INTERVENTIONS:
Drug: Tafasitamab — Given IV
  Other Names: MOR208
Drug: Lenalidomide — Given Orally
  Other Names: Revlimid

SUMMARY:
This is a single arm open-label multicenter phase I/II investigation of combination lenalidomide/Tafasitamab in patients with relapsed central nervous system (CNS) lymphoma. This is the first study to examine a naked anti-CD19 monoclonal antibody in relapsed CNS lymphoma patients as well as the combination of anti-CD19 antibody plus an Immunomodulatory imide drugs (IMiDs) in CNS lymphomas. This study will also test the novel hypothesis that Tafasitamab enhances blood-brain barrier permeability, a potential property that could have broad clinical implications.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) and recommended phase 2 dose (RP2D) of lenalidomide in combination with Tafasitamab in patients with relapsed central nervous system (CNS) lymphoma (Phase 1).

II. To evaluate the clinical benefit rate of Tafasitamab in combination with lenalidomide in relapsed CNS lymphoma (Phase 2).

SECONDARY OBJECTIVES:

I. To describe the toxicities of Tafasitamab in combination with lenalidomide in relapsed CNS lymphoma.

II. To describe the efficacy of Tafasitamab in combination with lenalidomide in relapsed CNS lymphoma.

EXPLORATORY OBJECTIVES:

I. To obtain pilot information about cerebral spinal fluid (CSF) penetration of Tafasitamab as well as CSF partition coefficient of lenalidomide in combination with Tafasitamab to evaluate possibility that Tafasitamab enhances CSF penetration of lenalidomide to an extent greater than CSF/plasma partition coefficient of lenalidomide which was 20% at 15 and 20 milligram (mg) dose levels.

II. To evaluate the relationship between tumor mutational profile and response to Tafasitamab plus lenalidomide, via whole exome sequencing of diagnostic specimens.

II. To evaluate change in immune cell phenotypes in CSF and blood in patients via flow-cytometry of natural killer (NK) cell, T-cells and CSF monocytes/macrophages in patients treated with combination Tafasitamab plus lenalidomide.

IV. To evaluate the relationship between CSF cytokine microenvironment such as Interleukin-10 (IL-10), Chemokine ligand 13 (CXCL13), etc. as well as CSF metabolites, including energy metabolites and neurotransmitters, and response to combination Tafasitamab plus lenalidomide Tafasitamab, PFS, OS, and neurocognitive endpoints.

V. To test the hypothesis that Tafasitamab in combination with lenalidomide impacts blood-brain barrier permeability associated with CNS lymphoma lesions, as assessed by albumin levels and MRI vascular permeability imaging metrics.

VI. To explore the correlation between immune cell subsets and response and/or resistance to lenalidomide/Tafasitamab.

VII. To evaluate the relationship between Minimal Residual Disease status (MRD) and response and PFS using either circulating tumor DNA or Clonoseq technologies.

STUDY DESIGN:

This is a single arm open-label multicenter phase I/II investigation of combination lenalidomide/Tafasitamab in patients with relapsed CNS lymphoma.During the phase 1 portion of the study, the investigators will examine three dose levels of Lenalidomide (10mg, 15mg and 20mg) in combination with Tafasitamab at a dose of 12 mg/kg. After MTD/RP2D is determined during phase 1, the phase 2 portion of the study will begin enrollment to the established dose.

Participants will be followed for AEs 90 days after last dose/decision to discontinue treatment, or new treatments are administered and followed for overall survival/disease status for up to 1 year after last dose. Participants may continue study treatment until disease progression.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must have relapsed primary or secondary CNS lymphoma, diffuse large B-cell lymphoma (DLBCL) type, based on radiographic, ophthalmologic, or CSF criteria (evidence of malignant cells based on CSF studies: cytospin/cytology and flow-cytometry).

   1. Concomitant systemic lymphoma as well as transformation from follicular lymphoma and/or Chronic lymphocytic leukemia (CLL) to an aggressive B-cell histology is allowed.
   2. Participants are eligible with disease in each CNS compartment: brain, leptomeninges/CSF and intraocular compartment.
2. Age >= 18 years.
3. Anticipated survival > 2 months, as determined by the investigator.
4. Eastern Cooperative Oncology Group (ECOG) performance status <=1 (Karnofsky performance status >= 70%)
5. Demonstrates adequate organ function as defined below:

   1. Absolute neutrophil count (ANC) ≥ 1.5 X 10^9/ L (1,500/ microliter (mcL), growth factors permitted).
   2. Platelets >= 50 X 10^9 / L (50,000/ mcL, platelet transfusion independent).
   3. Total bilirubin <= 1.5 x institutional upper limit of normal,unless elevated due to Gilbert's syndrome.
   4. Aspartate aminotransferase (AST)/serum glutamic-oxaloacetic transaminase (SGOT) <=3 X institutional upper limit of normal.
   5. Alanine aminotransferase (ALT)/serum glutamic-pyruvic transaminase (SGPT) <=3 X institutional upper limit of normal.

   d. Creatinine clearance (CrCl, calculated) >= 60 mL/min/1.73 m^2, calculated using the Cockcroft-Gault equation. CrCl > 60 mL/min/1.73 m2 is requisite for eligibility for the phase I dose-escalation phase of the study.
6. Ability to understand and the willingness to sign a written informed consent document.
7. For participants with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated. If a HBV test comes up positive due to Intravenous immunoglobulin (IVIG) and the participant has no prior history of HBV, then perform a HBV PCR to confirm.

   undetectable disease.
8. Individuals with a history of hepatitis C virus (HCV) infection must have been treated and cured. For individuals with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load.
9. Individuals with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
10. The effects of the study drugs on the developing human fetus are unknown. For this reason, and because the teratogenic effect of lenalidomide in humans cannot be ruled out, females of child-bearing potential (FCBP) and men must agree to use adequate contraception. FCBP must agree to undergo pregnancy testing as required in the study protocol. Should a woman become pregnant or suspect they are pregnant while their partner is participating in this study, they should inform her treating physician immediately.
11. Prior Therapies

    1. Participants with CNS lymphoma involving the brain parenchyma must have received at least one prior systemic therapy.
    2. Participants with secondary CNS lymphoma must have received prior CNS-directed treatment.
    3. There is no limit in terms of prior lines of therapy received. Patients may have progressed after prior treatment with IMiD's (including lenalidomide, pomalidomide and CC122), patients may have had prior rituximab or other anti-CD20 based therapy as well as autologous and allogeneic stem cell transplant. Patients who progress after prior stem cell transplant are immediately eligible whereas patients that progress after anti-CD19-based therapy including CAR-T based therapy are not eligible.
12. Recipients of prior hematopoietic stem cell transplant are eligible as long as the following criteria are met:

    1. Absence of graft versus host disease.
    2. Discontinuation of systemic immunosuppressant therapy.

Exclusion Criteria:

1. Has received systemic anti-cancer therapies within 2 weeks of first dose, radiation within 1 week, antibody therapy within 4 weeks.
2. Has not recovered from adverse events due to prior anti-cancer therapy to ≤ grade 1 or baseline (other than alopecia).
3. Is currently receiving any other investigational agents.
4. Has participated in a study of an investigational product and received study treatment or used an investigational device within four weeks of the first dose of treatment.
5. Has a history of HIV infection.
6. Has CNS post-transplant lymphoproliferative disease (PTLD).
7. Has known hypersensitivity to lenalidomide or Tafasitamab.
8. Pregnant women and women of child-bearing potential who will not using an effective method of birth control (detailed in Appendix 3) are excluded from this study because the study drugs have potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with lenalidomide and/or Tafasitamab, breastfeeding should be discontinued if the mother is treated with study drugs.
9. Prior receipt of anti-CD19 based therapy including anti-CD19, Chimeric antigen receptor T cells (CAR-T) therapy is an exclusion criteria.
10. Has any significant medical condition or comorbidity that could compromise patient safety (e.g., uncontrolled serious infection).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2022-06-08 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with dose limiting toxicities (DLTs) (Phase 1) | Up to 1 cycle (1 cycle is equal to 28 days)
  Toxicities will be classified using the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. The DLT will be based on the tolerability observed during the first cycle. In order for a patient to be assessed for DLT, they must receive at least 75% of lenalidomide dose (16 of the planned 21 days of lenalidomide administration). The maximum tolerated dose of lenalidomide/Tafasitamab will be the highest dose at which fewer than one-third of patients experience dose limiting toxicity. If multiple toxicities are seen, the presence of dose limiting toxicity should be based on the most severe toxicity experienced.
Maximum Tolerated Dose (MTD) (Phase 1) | Up to 1 cycle (1 cycle is equal to 28 days)
  The MTD is the highest dose at which no more than one instance of a DLT is observed among 6 participants treated.
Recommended Phase 2 Dose (RP2D) (Phase1) | Up to 1 cycle (1 cycle is equal to 28 days)
  The RP2D is the dose at which the Phase 2 portion of the study will begin enrolling. RP2D will be determined based on all data including available pharmacokinetics (PK), pharmacodynamic (PD), target engagement, efficacy, safety and tolerability data collected during Phase 1
Percentage of participants with demonstrated Clinical Benefit Rate (CBR) (Phase 2) | Up to 3 months
  Response to the combination lenalidomide/Tafasitamab treatment is defined as achieving clinical benefit better at three months restaging. That is overall tumor shrinkage within three months of treatment initiation or stable disease at three months restaging. Response criteria will be graded using the Cytologic Response Criteria, Neurologic Response Criteria, and Radiographic Response Criteria developed by the International Workshop to Standardize Baseline Evaluation and Response Criteria in Primary CNS Lymphoma The response rate is defined as the proportion of study participants meeting the definition of response in Efficacy Analysis Set (EAS). Response rate will be summarized by percentage, along with the corresponding exact 95% confidence intervals (CIs).

SECONDARY OUTCOMES:
Proportion of participants with Treatment-Related Adverse Events | Up to 90 days
  Serious adverse events, adverse events which are >=Grade 3, and adverse events resulting in discontinuation of treatment, withdrawal from the study, and deaths on-study will be used to determine the proportion of participants with treatment-related adverse events. Analyses will be performed based on the safety population.
Median Progression-free survival (PFS) (Phase 2) | Up to 1 year
  PFS is defined as the duration from first dose to disease relapse, progression, or death, whichever occurs first. The censoring time for PFS is set to be last study assessment for progression, and will be descriptively analyzed using Kaplan-Meier methods
Median Overall Survival (OS) | Up to 1 year
  OS is defined as the duration from first dose to death. The censoring time for OS is set to be the last study contact. OS will be descriptively analyzed using Kaplan-Meier methods.

CONTACTS AND LOCATIONS:
Overall Officials: James Rubenstein, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No